CLINICAL TRIAL: NCT00002154
Title: Parallel Group, Placebo-Controlled, Tolerability and Safety Study of Thioctic Acid and Deprenyl in HIV Dementia
Brief Title: A Study of Thioctic Acid and Deprenyl in HIV-Infected Patients With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Dana Foundation (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 250A; 03-D95
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Cognitive Disorders; HIV Infections
Keywords: Drug Therapy, Combination; Cognition Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Thioctic Acid; Selegiline
MeSH Terms: conditions — Cognitive Dysfunction; HIV Infections; Cognition Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Thioctic Acid; Selegiline

INTERVENTIONS:
Drug: Thioctic acid
Drug: Selegiline hydrochloride

SUMMARY:
The purpose of this study is to see if it is safe and effective to give thioctic acid and deprenyl (selegiline hydrochloride), alone or in combination, to HIV-infected patients who have mild to moderate dementia (a decline in their mental abilities).

DETAILED DESCRIPTION:
Patients are randomized to receive thioctic acid alone, deprenyl alone, thioctic acid/deprenyl, or placebo alone for 10 weeks, after which all patients may receive active drug on an open-label basis. Patients must have seven clinic visits.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretrovirals provided dose has been stable for at least 6 weeks prior to study entry.

Patients must have:

* HIV seropositivity.
* Mild to moderate cognitive impairment (problems with short term memory, concentration, and feeling slowed down).
* No active opportunistic CNS infection.
* Ability to give informed consent.

Prior Medication:

Allowed:

* Prior antiretrovirals provided dose has been stable for at least the past 6 weeks.
* Prior thioctic acid or deprenyl.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Severe premorbid psychiatric illness including schizophrenia and major depression that would interfere with study compliance.
* CNS neoplasms.
* Any other clinically significant condition or laboratory abnormality that would preclude participation on study.
* Current participation in other drug studies.

Concurrent Medication:

Excluded:

* Chemotherapy for malignancy.

Patients with the following prior conditions are excluded:

* History of chronic neurological disorders such as serious head injury, documented stroke, multiple sclerosis, uncontrolled epilepsy, Tourette's syndrome, and other neurodegenerative processes such as Huntington's disease.
* Prior participation in this study.
* History of adverse reaction/allergy to thioctic acid or deprenyl.

Prior Medication:

Excluded:

* Other investigational drugs within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Columbia Univ, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York